CLINICAL TRIAL: NCT00595998
Title: Sensitivity and Specificity of the Home Macular Perimeter
Brief Title: Sensitivity and Specificity of the Home Macular Perimeter (HMP)
Acronym: HMP
Status: Completed | Type: Observational
Sponsor: Notal Vision Ltd. (Industry)
Responsible Party: Dr. Josef Ferenzc, Meir Medical center
Organization: Notal Vision Inc. (Industry)
Other Study IDs: HMP-SS1; MMC-0206-07
Record Dates: First submitted 2008-01-06; First posted 2008-01-16 (Estimated); Last update posted 2009-01-28 (Estimated); Status verified 2009-01

CONDITIONS: Age Related Macular Degeneration
Keywords: AMD, HMP, PHP
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- 1: newly onset CNV secondary to AMD
- 2: Intermediate AMD

SUMMARY:
The primary objective of this study is to estimate the sensitivity of the HMP test in identifying visual field functional defects in subjects with CNV secondary to AMD, and differentiate them from intermediate AMD subjects.

DETAILED DESCRIPTION:
It is a one encounter visit in which patients are enrolled and complete the study on the same day. This will allow recruiting and testing of patients with CNV which is a dynamic disease that is most often treated on that same day. Following enrollment, patients will go through an examiner supervised tutorial followed by a self-performed HMP examination. In addition patient will undergo an Amsler grid examination, biomicroscopy, color fundus photography and fluorescein angiography. The HMP output shall be a test result that can be within or outside normal limits. Inherent to the test are reliability criteria which help to determine if the patient performed the test reliably. These consist of false positive and false negative errors. All criteria for normal limits and reliable performance are set prior to study initiation. The outcome measures for the study are the sensitivity in identifying visual functional defects in patients with CNV.

ELIGIBILITY:
Inclusion Criteria:

* Capable and willing to sign a consent form and participate in the study
* subjects with AMD related lesions: New onset (up to 60 days) non-treated CNV or Intermediate AMD patients (defined as the presence of at least one large drusen or more than 20 medium size drusen)
* Age >50 years
* VA with habitual correction >20/200 in study eye
* Familiar with computer usage

Exclusion Criteria:

* Evidence of macular disease other than AMD or glaucoma in the study eye
* Presence of any significant media opacity that precludes a clear view of the macular area as identified in the study eye by biomicroscopy, CFP, or FA
* Any non-macular related ocular surgery performed within 3 months prior to study entry in the targeted eye
* Inability to tolerate intravenous FA
* GA in the study eye
* Participation in another study with the exclusion of AREDS study

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The study population will include 30 subjects suspected to have newly onset CNV secondary to AMD in at least one eye, or Intermediate AMD in at least one eye, and who consent to participate in the study.
Sampling Method: Probability Sample
Enrollment: 42 (Actual)
Dates: Start 2008-01; Primary Completion 2008-09 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
estimate the sensitivity of the HMP test in identifying visual field functional defects in subjects with CNV secondary to AMD and differentiate them from intermediate AMD subjects. | 1 Month

CONTACTS AND LOCATIONS:
Overall Officials: Josef Mr Ferenzc, MD, Principal Investigator — Meir Medical Center
Locations (1):
- Meir Medical Center, Kfar Saba, Israel

REFERENCES:
- See also: Sponsor Site — http://www.notalvision.com